CLINICAL TRIAL: NCT01164072
Title: Randomised Controlled Trial Investigating the Efficacy and Safety of an Electronic Nicotine Delivery Device (E-Cigarette) in Smokers
Brief Title: Efficacy and Safety of an Electronic Nicotine Delivery Device (E-Cigarette)
Status: Completed | Type: Observational
Sponsor: Universita degli Studi di Catania (Other)
Collaborators: Lega Italiana Anti Fumo (Other); Arbi Group Srl (Industry)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor of Internal medicine, Universita degli Studi di Catania
Other Study IDs: CAT01/10
Record Dates: First submitted 2010-07-06; First posted 2010-07-16 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Smokers; Smoking Cessation
Keywords: electronic cigarette; nicotine; smoking cessation; smoking reduction
MeSH Terms: conditions — Smoking Cessation; Vaping; Smoking Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIGH NICOTINE: Well characterized group of 100 regular smokers experimenting the E-Cigarette loaded with 7.2 mg nicotine cartridges (high nicotine group).

SUMMARY:
The study's major aim is to investigate the ability of a commercial Electronic Nicotine Delivery Device (E-Cigarette) to induce long-term smoking reduction/abstinence in smokers unwilling to quit. Secondary aims are to investigate changes in withdrawal symptoms and cravings and to examine whether concomitant use of the E-Cigarette and smoking is safe.

The study will monitor smoking reduction/abstinence effects, changes in withdrawal symptoms, and adverse events of a currently marketed device in Italy ("Categoria" electronic cigarette - "ORIGINAL" 7.2 mg nicotine cartridges).

The primary hypothesis is that the E-Cigarette is a safe device that allows smoking reduction or abstinence in smokers possibly by suppressing withdrawal symptoms and cravings.

DETAILED DESCRIPTION:
The electronic cigarette (E-Cigarette) is an electronic nicotine delivery systems designed for the purpose of nicotine delivery to the respiratory system where nor tobacco nor combustion are necessary for its operation. For these reasons, it is possible that this product may be safer than cigarettes. Marketing claims also include that they can be useful smoking cessation aids. Although E-Cigarette may produce lung delivery of nicotine similar to that of tobacco cigarettes and reproduces the gesture component associated with tobacco smoking, very little is known about the effect of E-Cigarette on the smoking habits of regular tobacco smokers.

Therefore, we designed a prospective observational study consisting of 8 office-based visits (a baseline visit and a 2, 4, 6, 8, 10, and 12-weeks and a final visit at 24-weeks) to monitor possible modifications in the smoking habits of a group of well characterized regular smokers experimenting the e-cigarette focusing on long-term smoking reduction/abstinence, changes in withdrawal symptoms/cravings and adverse events.

Specifically, 100 smokers will be given "Categoria" electronic cigarette loaded with "ORIGINAL" 7.2 mg nicotine cartridges and followed up for a total of 24 weeks.

ELIGIBILITY:
Inclusion Criteria: healthy smokers unwilling to quit, between 18 and 60 years of age. They should report a cigarette intake of ≥ 15 cig/day for at least 5 years. At screening they must provide a CO level of ≥ 15 ppm and an FTND ≥ 5.

Exclusion Criteria: alcohol and illicit drug use, breastfeeding, or pregnancy. Individuals who report current attempts to quit smoking and previous experience with electronic cigarettes will be also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Regular smokers from Catania in Italy recruited following the placement of an advertisement in a local newspaper.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Sustained 50% reduction in the number of cigarettes smoked per day at week-12 from baseline | week-12
  50% reduction in the number of cigarettes smoked per day documented at each study visit (week-2, -4, -6, -8, -10, and -12)
Sustained smoking abstinence at week-12 | week 12
  Sustained smoking abstinence at week-12, defined as complete abstinence from tobacco smoking (not even a puff) for the 14 days period prior to week-12 study visit; exhaled CO levels will be measured to objectively verify smoking status.

SECONDARY OUTCOMES:
Sustained 80% reduction in the number of cigarettes smoked per day at week-12 from baseline | week-12
  80% reduction in the number of cigarettes smoked per day documented at each study visit (week-2, -4, -6, -8, -10, and -12)
Sustained smoking abstinence at week-24 | week 24
  Sustained smoking abstinence at week-24, defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to week-24 study visit; exhaled CO levels will be measured to objectively verify smoking status.
Sustained 50% reduction in the number of cigarettes smoked per day at week-24 from baseline | week-24
  50% reduction in the number of cigarettes smoked per day documented at each study visit (week-2, -4, -6, -8, -10, -12 and -24)
Sustained 80% reduction in the number of cigarettes smoked per day at week-24 from baseline | week-24
  50% reduction in the number of cigarettes smoked per day documented at each study visit (week-2, -4, -6, -8, -10, -12 and -24)
Withdrawal suppression (by MNWS) | 24 wks
Cravings reduction (by VAS) | 24 wks
Reported adverse events rate from baseline | 24 wks

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Polosa, MD, PhD, Principal Investigator — Università di Catania
Locations (1):
- Dipartimento di Medicina Interna e Specialistica; Centro per la Prevenzione e Cura del Tabagismo (CPCT), Catania, Italy

REFERENCES:
- [Derived] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093